CLINICAL TRIAL: NCT07212803
Title: Evaluation of Energy Drinks on Electrocardiographic Parameters: A Randomized, Double Blind, Controlled, Crossover, Proof-of-concept Study
Brief Title: Effects of Energy Drinks on Cardiovascular Endpoints
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Principal Investigator, Sachin Shah, Professor of Pharmacy Practice, University of the Pacific
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB2025-207
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Safety After Oral Intake
Keywords: Energy Drinks
MeSH Terms: interventions — Moxifloxacin; Caffeine; Control Groups; Taurine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Controlled, Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase A: Energy Drink A + Placebo (Experimental): Energy Drink A (320 mg caffeine) consumed with placebo capsule
  Interventions: Dietary Supplement: Energy Drink A + Placebo Capsule
- Phase A: Placebo Drink + Moxifloxacin (Active Comparator): Placebo drink with 400 mg moxifloxacin capsule
  Interventions: Drug: Placebo Drink + Moxifloxacin Capsule
- Phase A: Placebo Drink + Caffeine (Active Comparator): Placebo drink with 320 mg caffeine capsule
  Interventions: Dietary Supplement: Placebo Drink + Caffeine Capsule
- Phase A: Placebo Drink + Placebo Capsule (Placebo Comparator): Placebo drink with Placebo capsule
  Interventions: Other: Placebo Drink + Placebo Capsule
- Phase B: Energy Drink B (Experimental): Energy Drink B (320 mg caffeine)
  Interventions: Dietary Supplement: Energy Drink B
- Phase B: Control + Taurine (Experimental): Control product with 4000 mg taurine powder
  Interventions: Dietary Supplement: Control Product + Taurine
- Phase B: Control + Caffeine + Taurine (Experimental): Control product with 320 mg caffeine + 4000 mg taurine powder
  Interventions: Dietary Supplement: Control Product + Caffeine + Taurine
- Phase B: Lower Dose Energy Drink A (Experimental): Energy Drink A (189 mg caffeine)
  Interventions: Dietary Supplement: Lower Dose Energy Drink A

INTERVENTIONS:
Dietary Supplement: Energy Drink A + Placebo Capsule — 1000 mL caffeine- and taurine-containing commercially available beverage (Formula A) consumed with placebo capsule
  Arms: Phase A: Energy Drink A + Placebo
Drug: Placebo Drink + Moxifloxacin Capsule — Placebo drink with 400 mg moxifloxacin capsule
  Arms: Phase A: Placebo Drink + Moxifloxacin
Dietary Supplement: Placebo Drink + Caffeine Capsule — Placebo drink with 320 mg caffeine capsule
  Arms: Phase A: Placebo Drink + Caffeine
Other: Placebo Drink + Placebo Capsule — Placebo drink with placebo capsule
  Arms: Phase A: Placebo Drink + Placebo Capsule
Dietary Supplement: Energy Drink B — 568 mL caffeine- and taurine-containing commercially available beverage (Formula B)
  Arms: Phase B: Energy Drink B
Dietary Supplement: Control Product + Taurine — Control product with 4000 mg taurine powder
  Arms: Phase B: Control + Taurine
Dietary Supplement: Control Product + Caffeine + Taurine — Control product with 320 mg caffeine + 4000 mg taurine powder
  Arms: Phase B: Control + Caffeine + Taurine
Dietary Supplement: Lower Dose Energy Drink A — 591 mL caffeine- and taurine-containing commercially available beverage (Formula A)
  Arms: Phase B: Lower Dose Energy Drink A

SUMMARY:
This is a clinical trial looking at the impact of energy drinks on heart related parameters. The study will enroll 3 participants who will be exposed to 8 different interventions.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled, crossover, proof-of-concept trial designed to examine how energy drinks affect heart rhythm and other health measures in healthy adults aged 18 to 40. This study investigates the cardiovascular safety of energy drinks by examining their effects on electrocardiographic parameters, with a specific focus on the QTc interval.

The protocol consists of two phases conducted with 3 healthy volunteers. Phase A (Visits 1-4) evaluates four interventions: 1) energy drink A 2) moxifloxacin 3) caffeine 4) placebo.

Phase B (Visits 5-8) evaluates four interventions: 1) energy drink B 2) taurine 3) caffeine + taurine 4) lower dose energy drink A.

After an overnight fast participants will consume the study intervention within a 30 minute period. Over the next 4 hours, the electrocardiogram, blood pressure, hemodynamics, glucose, endothelial function, and side effects will be monitored. Participants maintain minimal physical activity during this period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults 18-40 years of age
* Female participants of child-bearing potential must have a negative pregnancy test at the baseline visit
* Participants must be willing to refrain from caffeine and alcohol use 72 hours prior to sessions on study days
* Participants must be willing and able to: (1.) Consume up to 1 liter of fluid within a 30-minute period per visit (2.) Swallow a single large capsule per visit
* Participants must be willing to fast 10 hours prior to sessions on study days (only water is allowed during the fasting and active study period)
* Participants must have active health insurance throughout the duration of the study

Exclusion Criteria:

* Have a corrected QT (QTc) interval greater than 450 milliseconds (ms) for males or greater than 470 milliseconds (ms) for females, determined during the baseline visit
* Presence of any known medical condition, confirmed through participant interview. Examples of these include but not limited to: Dyslipidemia, Thyroid disease, Diabetes, Recurrent headache, Any psychiatric condition or neurological disorder, History of alcohol or drug abuse, Past diagnosis or history of renal insufficiencies, Hepatic dysfunction, Electrolyte imbalances requiring hospitalization
* Presence of any known heart/cardiac diseases or conditions such as: Atrial Fibrillation, History of stroke or heart attack, Hypertension, Heart Failure, Vascular Disease, Family history/Active Long QT Syndrome, Coronary artery disease, Cardiomyopathy, Valvular heart disease, Ventricular arrhythmia, Congenital heart defect, Pericardial disease, Myocarditis
* Study physician recommendation for participant to not be enrolled.
* Are underweight (BMI<18.5 kg/m2, CDC 2024), have poor eating habits resulting in poor weight control, or have any factors that will put the participant at risk from fasting.
* Have any contraindications to the use of moxifloxacin, including a past medical history of myasthenia gravis, QT prolongation, or hypersensitivities and allergic reactions to moxifloxacin or any other fluoroquinolone antibiotics
* Pre-existing risk to tendinitis and tendon rupture, peripheral neuropathy, or central nervous system side effects
* Concurrent use of ANY medication taken daily including herbal products or supplements (daily basis is defined as greater than 2 days per week)
* Self-reported allergy to taurine
* Self-reported allergy to nuts (peanuts, pecans, cashews, etc.)
* Self-reported allergic reaction to the adhesive pads (electrodes, continuous glucose monitors, etc.)
* Fear of needle puncture
* Smokers using cigarettes, vaporized nicotine, or marijuana products currently or within the past month
* Current usage of any nicotine or tobacco products including but not limited to intranasal, sublingual, oral, or transdermal dosage forms
* Currently pregnant or breastfeeding
* Have a positive pregnancy test during the baseline visit
* Are currently enrolled in any other clinical study or have participated in another study within the last 30 days
* Non-English speaking/reading individuals will be excluded due to the unavailability of medically qualified translators throughout all study procedures
* If the candidate does not sign the informed consent document

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Corrected QT Interval (QTc) in Milliseconds (ms) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  QTc interval will be calculated using both Bazett's and Fridericia's correction formulas assessed via 12-lead ECG.

SECONDARY OUTCOMES:
Change from Baseline in QT Interval in Milliseconds (ms) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  As assessed via 12-lead ECG
Change from Baseline in RR Interval in Milliseconds (ms) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  As assessed via 12-lead ECG
Change from Baseline in PR Interval in Milliseconds (ms) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  As assessed via 12-lead ECG
Change from Baseline in QRS Duration in Milliseconds (ms) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  As assessed via 12-lead ECG
Change from Baseline in Systolic Blood Pressure (SBP) in Millimeters of Mercury (mmHg) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via a non-invasive automated blood pressure device
Change from Baseline in Diastolic Blood Pressure (DBP) in Millimeters of Mercury (mmHg) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via a non-invasive automated blood pressure device
Change from Baseline in Heart Rate (HR) in Beats Per Minute (BPM) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via non-invasive bioimpedance monitoring and/or 12-lead ECG
Change from Baseline in Cardiac Output (CO) in Liters Per Minute (L/min) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via non-invasive bioimpedance monitoring during Phase A only
Change from Baseline in Stroke Volume (SV) in Milliliters Per Beat (mL/beat) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via non-invasive bioimpedance monitoring during Phase A only
Change from Baseline in Interstitial Glucose Level (mg/dL) | Baseline, 30, 60, 90, 120, 150, 180, and 240 minutes post-intervention
  Assessed via a continuously worn arm sensor (Continuous Glucose Monitor, CGM) during Phase A only
Change from Baseline in Reactive Hyperemia Index (RHI) | Baseline, 120, and 240 minutes post-intervention
  A non-invasive, unitless measure of endothelial function assessed via peripheral arterial tonometry (EndoPAT) during Phase A only

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Pacific, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No